CLINICAL TRIAL: NCT04462783
Title: Feasibility of Self-monitoring and Patient Decision Support for Suspected COVID-19 Patients After Emergency Department Discharge
Brief Title: Emergency Department (ED) Self-Monitoring Pilot COVID-19
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Not funded
Sponsor: University of Michigan (Other)
Collaborators: Vironix Health Incorporated (Unknown)
Responsible Party: Principal Investigator, Kathleen Li, Adjunct Clinical Lecturer in Emergency Medicine, University of Michigan
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: HUM00181946
Record Dates: First submitted 2020-07-07; First posted 2020-07-08 (Actual); Last update posted 2021-07-01 (Actual); Status verified 2021-06

CONDITIONS: COVID; Covid-19; SARS-CoV 2
Keywords: coronavirus
MeSH Terms: conditions — COVID-19; Coronavirus Infections

STUDY DESIGN:
Intervention Model Description: Some patients will have pulse oximeters or be given one and provide data from these.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patient's symptom data without pulse oximeter (Experimental): Some patients may not be given a pulse oximeter to enter heart rate and O2 saturation into the CovidX application.
  Interventions: Other: Symptoms entered into the CovidX application
- Patient's symptom data with a pulse oximeter (Experimental): Some patients will be given (or may have) a pulse oximeter in order to enter heart rate and O2 saturation data into the CovidX application.
  Interventions: Other: Symptoms entered into the CovidX application

INTERVENTIONS:
Other: Symptoms entered into the CovidX application — Participants are asked to enter symptoms into the CovidX application at least daily for 30 days. Additionally, they will enter demographic information and some survey information will be collected.

SUMMARY:
This feasibility study is being conducted to understand how discharged emergency department patients who were tested for the SARS-CoV-2 virus (COVID-19) engage with a symptom-tracking web application. Study participants that are enrolled in the study will be asked to enter daily information about their health into the CovidX web application (app.). In addition, patients will answer questions regarding anxiety levels, use a pulse oximeter to record information (if you own one or are given one).

The investigators predict that participants will be able to engage with the CovidX web application over several days to weeks for the purposes of symptom tracking, and may have decreased anxiety over the study period.

ELIGIBILITY:
Inclusion Criteria:

* Reported symptoms of viral illness during ED encounter
* Tested for SARS-CoV-2 (COVID-19) during ED encounter
* Discharged home from the Emergency Department

Exclusion Criteria:

* Prisoners
* Residents of congregate living facilities who are already being monitored
* Baseline oxygen requirement
* Patients whose primary goals of care are palliative
* Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-06 (Estimated); Primary Completion 2021-11 (Estimated); Study Completion 2021-11 (Estimated)

PRIMARY OUTCOMES:
Change in the percent of participants using the CovidX web application (app) on 50% or greater of days | baseline, up to 30 days
Average compliance rate with daily symptom tracking by day 30 | Day 30
Recruitment rate | through study completion an average of 1 year
  The proportion of patients approached for the study who enroll

SECONDARY OUTCOMES:
Change in Patient-Reported Outcomes Measurement Information System (PROMIS) Anxiety short form 4a | completed at baseline (enrollment), up to 30 days
  The PROMIS Emotional Distress-Anxiety-Short Form 4a is a 4-item scale that assesses fear, anxiety, worry, and uneasiness. It uses a 5-point Likert scale (1 = never to 5 = always). Raw scores range from 4-20 with lower scores representing less endorsement of anxiety.
Change in Coronavirus Anxiety Scale | completed at baseline (enrollment), up to 30 days
  This is a 5- item questionnaire that assess anxiety related to the Coronavirus. Participants select from (0 = not at all to 4 = nearly every day over the last 2 weeks). The higher the total number the more anxiety.
CovidX web application usability and utility measured adapted by mHealth App Usability Questionnaire | 30 days
  The questionnaire is a series of 8 questions answered on a 1-7 Likert scale, with lower numbers indicating better usability. There are also 2 open-ended questions about why participants did or didn't like the application and other feedback is collected.
Differences in CovidX web application engagement between patients who do and do not receive a pulse oximeter | 30 days
  This will be measured by the compliance rates

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen Li, MD, Principal Investigator — University of Michigan